CLINICAL TRIAL: NCT05301543
Title: Behavioral Intervention to Reduce Sedative Use in Older Adults With Chronic Insomnia
Brief Title: Insomnia Behavioral Intervention Study
Acronym: IBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nalaka Gooneratne, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 849022
Record Dates: First submitted 2022-02-03; First posted 2022-03-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral approach 1 (Experimental): This includes sleep hygiene and other elements to serve as an experimental arm; subjects will receive a clinically proven therapeutic intervention.
  Interventions: Behavioral: Experimental: Behavioral approach 1
- Behavioral approach 2 (Active Comparator): This includes sleep hygiene and other elements to serve as an active comparator; subjects will receive a clinically proven therapeutic intervention.
  Interventions: Behavioral: Comparator: Behavioral approach 2

INTERVENTIONS:
Behavioral: Experimental: Behavioral approach 1 — Includes changing sleep habits and cognitions around sleep from a mental level
  Arms: Behavioral approach 1
Behavioral: Comparator: Behavioral approach 2 — Includes changing sleep habits and awarenes of sleep from a perception level
  Arms: Behavioral approach 2

SUMMARY:
This randomized pilot study (n=20) explores the effects of a behavioral intervention, that includes sleep hygiene improvements, in long-term users of sleeping pills, aiming to alleviate or stabilize symptoms of insomnia, monitor and decrease sleeping pill usage. Adherence will be monitored by an optional smartphone application.

DETAILED DESCRIPTION:
This randomized pilot study has a goal of enrolling 20 study participants. The investigators will examine the effects of a behavioral intervention, that includes sleep hygiene improvements such as regular sleep schedules, with assisted coaching support from the research team. Study participants are long-term users of sleeping pills. The goal is to improve or stabilizie insomnia symptoms and decrease sleeping pill usage. Study participant adherence will be monitored by an optional smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Age of 55-85
* Use of sleeping pill medication for sleep at least 3 nights a week
* Diagnosed with Chronic Insomnia by a physician
* Speaks English above a 6th-grade level
* Has access to a smartphone and/or smart tablet and can use it
* Has regular access to internet

Exclusion Criteria:

* Presence of major depression or other severe psychopathology (e.g., bipolar disorder, psychosis, alcohol/substance abuse, etc.)
* Presence of an acute or severe medical condition which, in the opinion of the research team, would interfere with the study participant's ability to participate in the research study, such as an acute heart attack, recent severe trauma, etc.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Sleep Pill Dosage | 28-day follow-up
  We will monitor changes in participants' sleep pill total dosage taken over one week using the sleep diary (which includes a daily question regarding sleeping pills used that night). The usage reduction will be calculated as a percent (total weekly usage at end of study divided by total weekly usage during the baseline week).

SECONDARY OUTCOMES:
Sleep Efficiency | 28-day follow-up
  Sleep efficiency which will be calculated using information from the sleep diary (logged daily from day 0 until day 28).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No